CLINICAL TRIAL: NCT06019143
Title: GoalNav® Clinic Module - Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ardea Outcomes (Other)
Collaborators: National Research Council, Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GoalNavRCC2023
Record Dates: First submitted 2023-08-09; First posted 2023-08-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: Eligible participants were sequentially assigned to inventory or no-inventory arms in parallel for the duration of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Inventory (Experimental): Goal Attainment Scaling (GAS) with goal inventory
  Interventions: Behavioral: Goal Attainment Scaling (GAS) with a goal inventory
- Arm B - No Inventory (Active Comparator): Goal Attainment Scaling (GAS) without goal inventory
  Interventions: Behavioral: Goal Attainment Scaling (GAS) without inventory

INTERVENTIONS:
Behavioral: Goal Attainment Scaling (GAS) with a goal inventory — Goal Attainment Scaling (GAS) with a goal inventory (list of common goals) as a behavioral interventional tool
  Arms: Arm A - Inventory
Behavioral: Goal Attainment Scaling (GAS) without inventory — Goal Attainment Scaling (GAS) without a goal inventory (list of common goals) as a behavioral interventional tool
  Arms: Arm B - No Inventory

SUMMARY:
This is a pilot study to test the feasibility of GoalNav® Clinic, an Electronic Data Capture platform which is specifically designed to collect data on patient goals, live in a clinical setting.

DETAILED DESCRIPTION:
Goal Attainment Scaling (GAS) is an individualized outcome measure that quantifies the effects of an intervention based on personalized goals.

Ardea Outcomes has developed an electronic data capture system called GoalNav® Clinic that is designed to capture GAS data (individual goals) in addition to other outcome measures that is useful to the doctor such as assessment information, patient demographics, cognitive status, etc..

With the help of a study doctor and/or a member of the research team trained in the process of conducting GAS interviews, patients and/or care partners set goals that are meaningful and relevant to them or their loved one's condition. Goals are then followed up in three months, and ratings are provided by the GAS interviewer and patient and/or care partner.

ELIGIBILITY:
Inclusion Criteria:

* a new or returning patient who has been referred and has a pre-scheduled appointment to the study doctor's clinic for a geriatric assessment
* of any age, with or without a disease diagnosis/memory complaint
* the patient is accompanied by a family member or friend who is willing to participate
* the patient and/or their care partner must be able to respond to questions in English
* the patient and their care partner give informed consent

Exclusion Criteria:

* the patient does not have a family member or friend who is willing to participate
* neither the patient nor their care partner can respond to questions in English
* either or both the patient and care partner decline to provide informed consent
* the study doctor deems that the patient and/or care partner is not suitable for the study
* either the patient or their care partner indicates on the informed consent form that they do not wish to be contacted by email or by telephone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Goal Setting Survey | 4 months
  The goal setting survey includes multiple choice, Likert type and open-ended questions with respect to the feasibility and acceptability of Goal Attainment Scaling. The questions focus on the impressions and experiences of patients and care partners (in Arm A and Arm B), and the study doctors when conducting interviews using GoalNav® EDC with and without goal inventory. The percentage of participants agreeing with statements with respect to ease of use, time commitment, etc. will be the unit of measurement. The answers to the open-ended questions will also be qualitatively analyzed.

SECONDARY OUTCOMES:
GAS Interviewer Individual Qualitative Interview | 4 months
  The one-hour qualitative interview with GAS interviewers will include questions such as
  * did GAS interviewers use the goal inventory for participants in Arm B (no goal inventory)?
  * was there a difference between Arm A and Arm B in the goal setting process?
  * was there a difference between Arm A and Arm B in goal quality?
  * did patients and care partners in Arm B find it difficult to identify challenges or goal areas without sufficient prompts?

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Kelly-Wiggins, MD, Principal Investigator — Nova Scotial Health
Locations (1):
- Geriatric Medicine & Memory Disability Clinic, Cape Breton Regional Hospital, Cape Breton, Nova Scotia, Canada

REFERENCES:
- [Background] Kiresuk TJ, Sherman RE. Goal attainment scaling: A general method for evaluating comprehensive community mental health programs. Community Ment Health J. 1968 Dec;4(6):443-53. doi: 10.1007/BF01530764. PMID 24185570